CLINICAL TRIAL: NCT00339079
Title: Treatment of Hypochondriasis With CBT and/or SSRI
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Arthur Joseph Barsky III,M.D., Vice Chair for Psychiatric Research, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01MH071688 (NIH); R01MH071688 (NIH)
Record Dates: First submitted 2006-06-16; First posted 2006-06-20 (Estimated); Results first posted 2017-03-03 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-03

CONDITIONS: Hypochondriasis
MeSH Terms: conditions — Hypochondriasis | interventions — Fluoxetine; olanzapine-fluoxetine combination; Cognitive Behavioral Therapy; Palliative Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cognitive Behavioral Therapy (CBT) (Experimental): Patients in this arm only received Cognitive Behavioral Therapy (CBT). Six, 60 minute weekly sessions were followed by 4 bi-weekly sessions and 3 monthly booster sessions.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)
- Placebo (Placebo Comparator): Patients only received placebo pills accompanied by medication management supportive therapy; including non-specific encouragement, support and explanation similar to that provide in a physician's office.
  Interventions: Other: Supportive Therapy; Drug: Placebo
- Fluoxetine (Experimental): Patients only received the SSRI Fluoxetine. Medication was adminstered on a fixed-flexible dosing regimen, beginning at 10mg/day for 2 weeks, then 20 mg/day for 2 weeks, 40 mg/day for two weeks, 60 mg/day for 2 weeks, and 80 mg/day (the target dose) thereafter. This was accompanied by medication management supportive therapy; including non-specific encouragement, support and explanation similar to that provide in a physician's office.
  Interventions: Drug: Fluoxetine; Other: Supportive Therapy
- Combined CBT and Fluoxetine (Experimental): Patients in this arm received both CBT and the fluoxetine medication. Both interventions were administered in the same way as when adminstered alone in the other arms.
  Interventions: Drug: Fluoxetine; Behavioral: Cognitive Behavioral Therapy (CBT)

INTERVENTIONS:
Drug: Fluoxetine — Each patient will receive fluoxetine in 10 or 20 mg pills given according to the following schedule: 10 mg/day for two weeks, 20 mg/day for two weeks, 40 mg/day for two weeks, 60 mg/day for two weeks, and 80 mg/day thereafter. The maximum dose for patients who are age 60 or older will be 60 mg/day. The study psychiatrist will have the option of not increasing or lowering the dose if hypochondriacal symptoms have resolved nearly completely for the last two weeks or adverse effects thought to be due to fluoxetine have occurred.
  Other Names: Prozac; Prodep; Sarafem; Lovan; Symbyax; Fluctin
  Arms: Combined CBT and Fluoxetine; Fluoxetine
Behavioral: Cognitive Behavioral Therapy (CBT) — CBT is based upon the cognitive and perceptual model of hypochondriasis and incorporates established behavioral techniques. There will be six 60-minute individual sessions conducted at weekly intervals. Booster sessions of 20 to 30 minutes will be conducted at Weeks 8 and 12. The introduction of boosters will make the CBT alone and medication alone arms identical in length.
  Arms: Cognitive Behavioral Therapy (CBT); Combined CBT and Fluoxetine
Other: Supportive Therapy — The supportive therapy component of the treatment is similar to what might occur in a family physician's office. Participants will meet with the same psychiatrist throughout the study, who will offer general encouragement; review the participant's illness, physical symptoms and, adverse effects over the previous week; and monitor medication dosage accordingly. Patients will be seen at Weeks 1, 2, 3, 4, 6, 8, 10, and 12, for medication adjustment. Visits with the psychiatrist will last 30 minutes.
  Arms: Fluoxetine; Placebo
Drug: Placebo — Each patient will receive placebo in 10 or 20 mg pills given according to the following schedule: 10 mg/day for two weeks, 20 mg/day for two weeks, 40 mg/day for two weeks, 60 mg/day for two weeks, and 80 mg/day thereafter.
  Arms: Placebo

SUMMARY:
This study will compare the effectiveness of cognitive behavioral therapy, antidepressant medication, and a combination of the two for treating hypochondriasis.

DETAILED DESCRIPTION:
Hypochondriasis is one of the most difficult psychiatric disorders to treat. People with hypochondriasis believe that real or imagined physical symptoms are signs of serious illnesses, despite medical reassurance and other evidence to the contrary. Symptoms of the disorder include a preoccupation with fear of an illness; a persistent fear of having a serious illness, despite medical reassurance; and misinterpretation of symptoms. Some individuals with hypochondriasis recognize that their fear of having a serious illness may be excessive, unreasonable, or unfounded. Episodes of hypochondriasis usually last from months to years, with equally long periods of remission. Cognitive behavioral therapy (CBT) and the antidepressant drug fluoxetine (FLX) have both been shown to be effective treatments for hypochondriasis. However, the relative efficacy of a combined approach has yet to be determined. This study will compare the effectiveness of cognitive behavioral therapy, antidepressant medication, and a combination of the two for treating hypochondriasis.

Participants in this double-blind study will first report to the study site for two sessions to determine eligibility for participation. Eligible individuals will then be randomly assigned to receive one of the following four treatments for 12 weeks: CBT only; FLX only; CBT plus FLX; or a placebo pill. All participants receiving medication will also receive supportive therapy. Treatment response will be assessed at Week 12, and participants who have shown improvement will continue in the study for an additional 12 weeks. Participants who have not responded to treatment will be removed from the study and will receive open treatment. Participants assigned to receive medication or placebo will take medication once daily for the full 24 weeks. Participants assigned to CBT only or CBT plus FLX will receive CBT weekly for the first 8 weeks, then biweekly until Week 12, and then monthly until week 24. Outcomes will be assessed at study visits at Weeks 6, 12, 24, and 48, and over the phone at Week 36.

ELIGIBILITY:
Inclusion Criteria

* Meets DSM-IV criteria for hypochondriasis; ascertained by Structured Diagnosis for Hypochondriasis module of SCID-I, and meets a hypochondriasis severity rating of at least "moderate".
* Drug free for 6 weeks of all psychoactive or investigational medications (seven weeks for fluoxetine).
* Approval from treating physician if concomitant psychoactive medications need to be withdrawn prior to study participation.
* English fluency and literacy.

Exclusion Criteria

* Pregnant or nursing mothers and women of childbearing potential who are not taking adequate birth control precautions.
* Any of the following Axis I mental disorders: chronic pain syndrome, schizophrenia, schizoaffective disorder, delusional disorder, bipolar disorder, alcohol abuse or dependence disorder (current or within the last six months), or substance abuse or dependence disorder (current or within the last twelve months). Patients with other comorbid psychiatric disorders are eligible based on the following three criteria: hypochondriasis must be the predominant presenting disorder; patient can not have a major co-morbid psychiatric disorder rated as "severe" on the Clinical Global Impressions Scale (CGI Scale); and patients can not have a co-morbid psychiatric disorder that causes significant functional impairment (significant functional impairment will be defined as an impairment that interferes in a marked way with expected role functioning, vocational and/or interpersonal).
* Suicidality within the last 6 months as established by a score of 9 or more on the suicidality module of the MINI Plus.
* Symptom-contingent pending litigation, disability compensation, or workers' compensation proceedings
* Major medical illness expected to worsen significantly, lead to hospitalization, or likely to prove fatal in the next six months, established with the Cumulative Illness Rating Scale (CIRS); Stable, chronic medical illness is not an exclusion criterion
* Not able to withdraw from concomitant psychoactive medications or currently taking necessary other medication that might interact adversely with fluoxetine:
* Clinically important abnormalities in ECG, laboratory tests (including thyroid function) or physical examination. "Clinically important" abnormalities are those that signify a treatment intervention is needed or a medical abnormality has not been sufficiently addressed. Patients with medical problems that are stable and chronic are eligible, but patients with medical problems that are unstable, acute, or inadequately evaluated will be excluded. A current electrocardiogram is required for all patients with symptoms suggestive of cardiac disease, including chest pain, dyspnea, palpitations, or lightheadedness; if no current electrocardiogram exists, the study will obtain one.
* History of severe side effects associated with fluoxetine or noncompliance with prior CBT for hypochondriasis
* Previous adequate trial of either fluoxetine (eight weeks of which two weeks were at a minimum dose of 60 mg/day) or CBT for hypochondriasis (at least four sessions specifically targeting hypochondriacal symptoms) will be excluded, regardless of prior response. Inability to ambulate or mobility restrictions that prohibit frequent travel to the hospital for treatment and evaluation.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2006-06; Primary Completion 2011-05 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur J. Barsky, MD, Principal Investigator — Brigham and Women's Hospital and Harvard Medical School; Brian Fallon, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Columbia Medical Center, New York Psychiatric Institute, New York, New York

REFERENCES:
- [Background] Barsky AJ, Ahern DK. Cognitive behavior therapy for hypochondriasis: a randomized controlled trial. JAMA. 2004 Mar 24;291(12):1464-70. doi: 10.1001/jama.291.12.1464. PMID 15039413
- [Background] Barsky AJ, Wyshak G. Hypochondriasis and somatosensory amplification. Br J Psychiatry. 1990 Sep;157:404-9. doi: 10.1192/bjp.157.3.404. PMID 2245272
- [Background] Barsky AJ. A 37-year-old man with multiple somatic complaints. JAMA. 1997 Aug 27;278(8):673-9. No abstract available. PMID 9272901
- [Derived] Fallon BA, Ahern DK, Pavlicova M, Slavov I, Skritskya N, Barsky AJ. A Randomized Controlled Trial of Medication and Cognitive-Behavioral Therapy for Hypochondriasis. Am J Psychiatry. 2017 Aug 1;174(8):756-764. doi: 10.1176/appi.ajp.2017.16020189. Epub 2017 Jun 29. PMID 28659038
- [Derived] Scarella TM, Laferton JA, Ahern DK, Fallon BA, Barsky A. The Relationship of Hypochondriasis to Anxiety, Depressive, and Somatoform Disorders. Psychosomatics. 2016 Mar-Apr;57(2):200-7. doi: 10.1016/j.psym.2015.10.006. Epub 2015 Oct 23. PMID 26785798

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was from October 2003 to July 2008. Participants were recruited via advertisements to the general public (e.g., newspaper ads).
Period: Overall Study
Arm/Group | Cognitive Behavioral Therapy (CBT) | Placebo | Fluoxetine | Combined CBT and Fluoxetine
Started | 53 | 44 | 45 | 53
Completed | 20 | 21 | 27 | 29
Not Completed | 33 | 23 | 18 | 24

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Patients only received placebo pills
- Fluoxetine: Patients only received the SSRI Fluoxetine. Medication was adminstered on a fixed-flexible dosing regimen, beginning at 10mg/day for 2 weeks, then 20 mg/day for 2 weeks, 40 mg/day for two weeks, 60 mg/day for 2 weeks, and 80 mg/day (the target dose) thereafter.
- Combined CBT and Fluoxetine: Patients in this arm received both CBT and the fluoxetine medication. Both interventions were administered in the same way as when administered alone in the other arms.
- Total: Total of all reporting groups
Arm/Group | Cognitive Behavioral Therapy (CBT) | Placebo | Fluoxetine | Combined CBT and Fluoxetine | Total
Number analyzed (Participants) | 53 | 44 | 45 | 53 | 195
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (13.7) | 36.4 (12.9) | 43.1 (15.9) | 40.0 (14.3) | 39.7 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 15 | 25 | 21 | 85
  Male | 29 | 29 | 20 | 32 | 110
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 9 | 6 | 23
  Not Hispanic or Latino | 48 | 41 | 36 | 47 | 172
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: 25% Improvement on Both Whiteley Index and H-YBOCS-M
Description: Whitley index is a self-report measure of hypochondriasis H-YBOCS-M is an independent evaluator structured assessment of hypochondriasis
Time Frame: Measured at Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitive Behavioral Therapy (CBT) | Placebo | Fluoxetine | Combined CBT and Fluoxetine
Number analyzed (Participants) | 53 | 44 | 45 | 53
Participants | 21 | 13 | 20 | 25

2. Secondary Outcome: Columbia Heightened Illness Concern - Obsessive-Compulsive Scale
Description: The Columbia Heightened Illness Concern - Obsessive-Compulsive Scale was the name for an earlier version of the H-YBOCS-M. The H-YBOCS-M is an expanded version and has additional items not included in the Columbia Heightened Illness Concern OCS. We did not administer the CHIC-OCS to patients in this study.
Time Frame: Not measured
Groups:
- Fluoxetine: Patients received the SSRI Fluoxetine. Medication was adminstered on a fixed-flexible dosing regimen, beginning at 10mg/day for 2 weeks, then 20 mg/day for 2 weeks, 40 mg/day for two weeks, 60 mg/day for 2 weeks, and 80 mg/day (the target dose) thereafter. This was accompanied by medication management supportive therapy; including non-specific encouragement, support and explanation similar to that provide in a physician's office.
  Fluoxetine: Each patient will receive fluoxetine in 10 or 20 mg pills given according to the following schedule: 10 mg/day for two weeks, 20 mg/day for two weeks, 40 mg/day for two weeks, 60 mg/day for two weeks, and 80 mg/day thereafter. The maximum dose for patients who are age 60 or older will be 60 mg/day. The study psychiatrist will have the option of not increasing or lowering the dose if hypochondriacal symptoms have resolved nearly completely for the last two weeks or adverse effects thought to be due to fluoxetine have occurred.
  Supportiv
- Combined CBT and Fluoxetine: Patients arm received both CBT and the fluoxetine medication. Both interventions were administered in the same way as when adminstered alone in the other arms.
  Fluoxetine: Each patient will receive fluoxetine in 10 or 20 mg pills given according to the following schedule: 10 mg/day for two weeks, 20 mg/day for two weeks, 40 mg/day for two weeks, 60 mg/day for two weeks, and 80 mg/day thereafter. The maximum dose for patients who are age 60 or older will be 60 mg/day. The study psychiatrist will have the option of not increasing or lowering the dose if hypochondriacal symptoms have resolved nearly completely for the last two weeks or adverse effects thought to be due to fluoxetine have occurred.
  Cognitive Behavioral Therapy (CBT): CBT is based upon the cognitive and perceptual model of hypochondriasis and incorporates established behavioral techniques. There will be six 60-minute individual sessions conducted at weekly intervals. Booster sessions of 20 to 30 minutes wi
Arm/Group | Cognitive Behavioral Therapy (CBT) | Placebo | Fluoxetine | Combined CBT and Fluoxetine
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were continually collected and reported annually when the continuing review was submitted to the human research committee.
Arm/Group | Cognitive Behavioral Therapy (CBT) | Placebo | Fluoxetine | Combined CBT and Fluoxetine
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/44 | 0/45 | 0/53
Other Adverse Events (participants affected / at risk) | 0/53 | 1/44 | 0/45 | 0/53
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Behavioral Therapy (CBT) (N=53) | Placebo (N=44) | Fluoxetine (N=45) | Combined CBT and Fluoxetine (N=53)
Medication Switch (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — 1 subject was inadvertently switched from receiving the placebo, to which she had been randomly assigned, to receiving fluoxetine, the active study medication.

LIMITATIONS AND CAVEATS:
1) Limited generalizability since we studied volunteers not medical patients. 2) Sampling bias possible as many subjects sought CBT and were unwilling to take chance of being randomized to medication. 3) Relatively high rates of attrition.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No